CLINICAL TRIAL: NCT03702049
Title: Nurse-Led Community Health Worker Adherence Model in 3HP Delivery Among Homeless Adults at Risk for TB Infection and HIV
Acronym: 3HP-LTBI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Irvine (Other)
Collaborators: University of California, Los Angeles (Other); National Institute on Minority Health and Health Disparities (NIMHD) (NIH)
Responsible Party: Principal Investigator, Adeline Nyamathi, Founding Dean and Distinguished Professor, University of California, Irvine
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 20184698; R21MD012696 (NIH)
Record Dates: First submitted 2018-10-08; First posted 2018-10-10 (Actual); Results first posted 2024-04-18 (Actual); Last update posted 2024-04-18 (Actual); Status verified 2024-03

CONDITIONS: Latent Tuberculosis Infection
MeSH Terms: conditions — Latent Tuberculosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- RN/CHW TBI (Experimental): Nurse-led Community Health Worker TBI (RN/CHW TBI) program
  Interventions: Behavioral: Nurse-led Community Health Worker TBI (RN/CHW TBI) program

INTERVENTIONS:
Behavioral: Nurse-led Community Health Worker TBI (RN/CHW TBI) program — Homeless adults with TBI will be assigned to this program which includes culturally-sensitive education, case management, and directly observed therapy (DOT) delivery of medication among patients who have been prescribed 3HP (12 weeks treatment for latent TB infection) by a medical provider. For this research, 3HP will be delivered to homeless persons infected with TB on a weekly basis by CHW under the guidance of their RN. The RN/CHW team will also provide case management, including health education and referrals for social services.

SUMMARY:
Tuberculosis (TB) is the prototypical disease of poverty as it disproportionately affects marginalized and impoverished communities. In the US, TB rates are unacceptably high among homeless persons who have a 10-fold increase in TB incidence as compared to the general population. In California, the rate of TB is more than twice the national case rate and recent TB outbreaks have been alarming. Among persons with active TB disease, over 10% die during treatment, with mortality being even higher among homeless persons with TB. While TB can be prevented by treating TB infection (TBI) before it develops into infectious, symptomatic disease, individual factors such as high prevalence of psychosocial comorbidities, unstable housing and limited access to care have led to poor adherence and completion of TBI treatment among homeless persons.

Given the complex health disparity factors that affect TBI treatment adherence among homeless persons, this study will assess the feasibility of a theoretically-based novel model of care among persons with TBI and complex chronic illnesses. This study will evaluate an innovative, community-based intervention that addresses critical individual level factors which are potential mechanisms that underlie health disparities in completing TBI treatment among the predominantly minority homeless. The study hypothesis is that improving these conditions, and promoting health by focused screening for TBI, and early detection and treatment for these vulnerable adults will improve TB treatment completion and prevent future TB disease.

The proposed theoretically-based health promotion intervention focuses on: 1) completion of TBI treatment, 2) reducing substance use; 3) improving mental health; and 4) improving critical social determinants of TB risk (unstable housing and poor health care access) among homeless adults in the highest TB prevalence area in Los Angeles. A total of 76 homeless adults with TBI will receive this program which includes culturally-sensitive education, case management, and directly observed therapy (DOT) delivery of medication among patients who have been prescribed 3HP (12 weeks treatment for latent TB infection) by a medical provider. This study will determine whether this intervention can achieve higher completion rates than the 65% completion rate among homeless persons reported by previous TB programs.

DETAILED DESCRIPTION:
Tuberculosis (TB) is a global public health threat, which is driven by social factors, including poverty, inadequate housing, malnutrition, and substance use. In the United States (US), TB disproportionately impacts homeless populations. When compared to the general population, homeless persons have a 10-fold increase in TB incidence. Lack of stable housing and living in congregate settings are predisposing factors for TB Infection (TBI). Homeless persons who develop active TB disease are also at higher risk of death during TB treatment due to mental illness and substance use. Even one TB case among a homeless person can easily lead to widespread TB transmission due to crowded, poorly ventilated, and congregate living situations. Therefore, an extensive public health response is needed for each case of infectious TB disease that develops among homeless persons.

Given the significant public health impact of TB among homeless persons, development of effective interventions to prevent TB among homeless persons that are theoretically-based and advance science in the area of best adherence strategies to minimize these health disparities can lead to significant benefits for patients and further reduce the disparity in TB rates between homeless and housed persons. While adherence to traditional TBI treatment with 6 to 9 months of isoniazid (INH) has been dismal, over the last few years, a promising treatment option in form of a 12-dose combination therapy (3HP; rifapentine [RPT] plus isoniazid [INH]), delivered once weekly as directly observed therapy (DOT), has achieved treatment completion rates of 82%. However, homeless populations who are at high risk for TBI have complex, multi-dimensional barriers to TBI treatment adherence. Thus, TBI treatment programs in this population have yielded marginal results of 65% completion to date. Among homeless persons, health disparities are accentuated by additional barriers to TBI treatment adherence, including substance use, mental disorders, and unstable housing.

Given the complex factors that affect TBI treatment adherence among homeless persons, the research team developed a theoretically-based novel model of care that has been successfully investigated in other disadvantaged populations. This model involves understanding the behavioral, psychological, and environmental influences on health and developing culturally-tailored interventions to reduce health disparities, and promote health. By engaging nurses, physicians, and community health workers (CHW), the investigators have developed a team-based approach to better understand and support medication adherence by engaging individuals as active partners in managing their own health. This scientific contribution has the potential to be highly significant as new models of care are being proposed to improve timely entry, engagement and retention in care, and supportive services for homeless persons and other vulnerable populations affected by complex health disparities impacting treatment adherence. The pilot study builds on the investigators' extensive three decades of research with homeless persons in improving health, including TBI treatment adherence, HBV vaccination, and adherence to HIV therapy.

This study will assess the impact of the TBI program that the investigators have developed, as a single arm intervention study, among 76 eligible TBI homeless adults on completion of 3HP treatment, decrease in drug and alcohol use, improved access to care and mental health, and shelter stability. Completion of 3HP will be compared to a minimum standard completion rate of 65%. This small pilot will generate the effectiveness data for a future R01 application to evaluate the intervention in a definitive randomized-controlled trial (RCT).

ELIGIBILITY:
Inclusion Criteria:

* self-reported homeless adults (past six months);
* age 18 or older;
* willing to provide informed consent;
* positive for TBI
* reported current or recent substance use (past three years)

Exclusion Criteria:

* screened as having active TB or currently treated for TBI;
* history of treatment for active TB or TBI;
* a serum aspartate aminotransferase (AST) level of 3-5 times the upper limit of normal;
* HIV infected AND receiving antiretroviral therapy (as 3HP is not recommended yet in this group);
* not able to speak English or Spanish;
* testing pregnant (as 3HP is not recommended in this group); and
* judged to be cognitively impaired

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2019-01-24 (Actual); Primary Completion 2020-05-29 (Actual); Study Completion 2020-09-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Adeline M Nyamathi, PhD, Principal Investigator — University of California, Irvine
Locations (2):
- United States (2):
  - Los Angeles Christian Health Centers (LACHC), Los Angeles, California
  - Union Rescue Mission, Los Angeles, California

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Nyamathi A, Salem BE, Shin SS, Jones AA, Garfin DR, Yadav K, Chang AH, White K, Morisky D. Effect of a Nurse-Led Community Health Worker Intervention on Latent Tuberculosis Medication Completion Among Homeless Adults. Nurs Res. 2021 Nov-Dec 01;70(6):433-442. doi: 10.1097/NNR.0000000000000545. PMID 34380979

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 466 were screened. Of these, 250 were determined as not meeting inclusion criteria as follows: PPD negative (n=178); QFT negative (n=18); Previous LTBI tx completion (n=22); Moved out of state (n=2); CXR positive (n=1); HIV positive (n=1); Not homeless (n=8); Did not have mental illness, substance use or medical care while homeless (n=12); Not willing to take blood test (n=3); Not willing to take medication (n=5); Declined to participate (n=13); and Failed to return (n=153).
Groups:
- RN/CHW TBI: This is a single-arm trial with all participants assigned to receive the multi-component intervention, including the 3HP medication.
Period: Overall Study
Arm/Group | RN/CHW TBI
Started | 50
Completed | 45 (Of the 50 enrolled, one was asked to discontinue the medication per physician provider. Of the 49 who underwent analysis, 45 completed the medication (1 moved out of state and 3 were lost to follow-up.)
Not Completed | 5
Not completed — Lost to Follow-up | 4
Not completed — Physician Decision | 1

BASELINE CHARACTERISTICS:
Arm/Group | RN/CHW TBI
Number analyzed (Participants) | 50
Age, Continuous [Mean (Standard Deviation); unit: years] | 53.7 (12.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13
  Male | 37
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 21
  Not Hispanic or Latino | 29
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 4
  Asian | 2
  Native Hawaiian or Other Pacific Islander | 2
  Black or African American | 24
  White | 6
  More than one race | 12
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 50

OUTCOME MEASURES:

1. Primary Outcome: Completion of TBI Treatment
Description: Completion of TBI Treatment will be measured at 3 month follow-up by 90% completion of medication (at least 11/12 doses) consumed over a 12 week period
Time Frame: 3 months (12 weeks)
Population: Participants with 3 month follow-up visit completed
Measure: Count of Participants; unit: Participants
Arm/Group | RN/CHW TBI
Number analyzed (Participants) | 49
Participants | 45

2. Secondary Outcome: Drug Use
Description: Assessed by the drug items in the Texas Christian University (TCU) Screen V. Yes/No responses to substance dependency questions and the frequency of drug use based on a 5-point scale from 1 (never) to 5 (daily) will be assessed for each drug used. The total score ranges from 0 - 11; corresponding to the number of symptoms endorsed by the participant and the severity of SUD: mild disorder (2-3 points), moderate disorder (4-5 points), or severe disorder (6 or more points).
Time Frame: baseline, 3 and 6 months
Population: Participants who completed 6 months of follow-up
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | RN/CHW TBI
Number analyzed (Participants) | 45
score on a scale
  Baseline | 1.98 (3.02)
  3 month | 1.64 (2.84)
  6 month | 1.8 (3.47)
Statistical Analysis 1: Comparison: RN/CHW TBI; Change in score at 3 months; Test type: Other — Change in score at 3 months; p = 0.603, Mixed Models Analysis; Mean Difference (Final Values) = -0.24
Statistical Analysis 2: Comparison: RN/CHW TBI; 6 month outcome; Test type: Other — Change at 6 months; p = 0.805, Mixed Models Analysis; Mean Difference (Final Values) = -0.12

3. Secondary Outcome: Alcohol Use
Description: Assessed by the Alcohol items in the Texas Christian University (TCU) Screen V. Problematic use of alcohol was defined as self-identified as being a problem (TCU Item #12) or daily consumption.
Time Frame: baseline, 3 and 6 months
Population: Participants who completed 6 months of follow-up
Measure: Count of Participants; unit: Participants
Arm/Group | RN/CHW TBI
Number analyzed (Participants) | 45
Participants
  Baseline | 14
  3 month: number analyzed (Participants) | 44
  3 month | 11
  6 month: number analyzed (Participants) | 38
  6 month | 7
Statistical Analysis 1: Comparison: RN/CHW TBI; 3 month outcome; Test type: Other; p = 0.672, Regression, Logistic; Odds Ratio (OR) = 0.83, 95% CI 2-sided [0.39 to 1.79]
Statistical Analysis 2: Comparison: RN/CHW TBI; 6 month outcome; Test type: Other; p = 0.165, Regression, Logistic; Odds Ratio (OR) = 0.49, 95% CI 2-sided [0.18 to 1.34]

4. Secondary Outcome: Depression
Description: Depression will be assessed by the Center for Epidemiological Studies Short Depression Scale Revised (CESD-R-10) is a 10-item measure for depressive symptoms in the past week (endpoints 0=rarely or none of the time; 3=most of the time). Scale range 0-30, with greater values meaning worse depressive symptoms. Responses are summed.
Time Frame: baseline, 3 and 6 months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | RN/CHW TBI
Number analyzed (Participants) | 45
score on a scale
  Baseline | 9.11 (6.07)
  3 month | 8.84 (4.82)
  6 month | 9.4 (5.3)
Statistical Analysis 1: Comparison: RN/CHW TBI; 3 month outcome; Test type: Other; p = 0.719, Mixed Models Analysis; Mean Difference (Final Values) = -0.31
Statistical Analysis 2: Comparison: RN/CHW TBI; 6 month outcome; Test type: Other; p = 0.626, Mixed Models Analysis; Mean Difference (Final Values) = 0.43

5. Secondary Outcome: Health Care Access
Description: Health Care Access will include number of healthcare visits made
Time Frame: 3 and 6 months
Measure: Mean (Standard Deviation); unit: Visits
Arm/Group | RN/CHW TBI
Number analyzed (Participants) | 45
Visits
  3 month | 4.33 (2.27)
  6 month | 3.18 (2.66)
Statistical Analysis 1: Comparison: RN/CHW TBI; Test type: Other; p = 0.1668, t-test, 2 sided; Mean Difference (Final Values) = 0.83, 95% CI 2-sided [-0.36 to 2.03]

6. Secondary Outcome: Shelter Stability - Days Residing in the Shelter
Description: Shelter Factors: Staff will record the type of residence at baseline and follow-up. Shelter Stability will be assessed by the length of time in days residing in the shelter
Time Frame: 3 and 6 months
Measure: Mean (Standard Deviation); unit: days
Arm/Group | RN/CHW TBI
Number analyzed (Participants) | 45
days
  Baseline | 76.8 (59.9)
  3 month | 82 (16.8)
  6 month | 74.3 (24.6)
Statistical Analysis 1: Comparison: RN/CHW TBI; 3 month outcome; Test type: Other; p = 0.9198, t-test, 2 sided; Mean Difference (Final Values) = 1.5, 95% CI 2-sided [-29.6 to 32.7]
Statistical Analysis 2: Comparison: RN/CHW TBI; 6 month; Test type: Other; p = 0.5015, t-test, 2 sided; Mean Difference (Final Values) = 12.5, 95% CI 2-sided [-25.6 to 50.7]

ADVERSE EVENTS:
Time Frame: 3 months
Description: Adverse effects were typical side effects of the prescribed medication
Arm/Group | RN/CHW TBI
All-Cause Mortality (participants affected / at risk) | 0/50
Serious Adverse Events (participants affected / at risk) | 0/50
Other Adverse Events (participants affected / at risk) | 9/50
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | RN/CHW TBI (N=50)
Loss of apetite (Metabolism and nutrition disorders) | 3 (3)
Unexplained anorexia (Metabolism and nutrition disorders) | 3 (3)
Abdominal pain (Gastrointestinal disorders) | 3 (3)
Nausea (Gastrointestinal disorders) | 5 (5)
Easy Bruising or Bleeding (General disorders) | 3 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2024-01-02): https://cdn.clinicaltrials.gov/large-docs/49/NCT03702049/Prot_SAP_000.pdf